CLINICAL TRIAL: NCT04080232
Title: Study of Pulmonary MRI for the Diagnosis of Bronchiolitis Obliterans Syndrome After Allogeneic Stem Cell Transplantation
Acronym: IRM-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: SFGM-TC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/05
Record Dates: First submitted 2019-07-04; First posted 2019-09-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Bronchiolitis Obliterans
Keywords: lung MRI performance; UTE; quantification; oxygen transfer; Bronchiolitis Obliterans syndrome; allogeneic stem cell transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lung MRI (Experimental): lung MRI concordance as compared to chest CT-scan for the description of morphological abnormalities necessary for the diagnosis of BOS after HSCT. It will be evaluated using lung MRI performed after inclusion (D0) using a standardized procedure
  Interventions: Device: lung MRI

INTERVENTIONS:
Device: lung MRI — lung MRI (1.5T Siemens Aera) using the following sequences: 3D Fast gradient-echo pulse sequences with ultra-short echo time (UTE), acquisitions at end-inspiration breath hold, end-expiration breath hold, and free-breathing using an echonavigator positioned on the diaphragm, acquisitions using routine pulse sequences (SSFP, T2FSE) and the administration of oxygen during the MRI: O2 will be administered at 15L/min during 6 minutes.

SUMMARY:
Bronchiolitis Obliterans Syndrome (BOS) is a major complication of Hematopoietic Stem cell Transplantation (HSCT) occurring in the context of chronic GVHD and associated with a poor prognosis. The diagnosis of BOS is based on functional (Pulmonary Functional Tests) and morphological criteria (chest CT-scan). Early diagnosis of BOS represents an unmet need and would facilitate early therapeutic interventions. Lung MRI has been recently developed with new sequences facilitating morphological and functional lung analysis in various inflammatory contexts. The goal of this study is to compare the morphological performances of chest CT-scan and MRI

DETAILED DESCRIPTION:
Patients undergoing allogeneic stem cell transplantation may develop non-infectious respiratory complication related to chronic graft versus host disease and called bronchiolitis obliterans syndrome (BOS). The occurrence of BOS is associated with a decreased survival reaching 13% at 5 years (Dudek et al, BBMT 2003). Thus, screening and diagnosis of BOS appear as a priority of post-transplant patients monitoring, in order to begin early therapy if needed. To this end, patients undergo systematic and regular screening using pulmonary function tests (PFTs). In case of abnormal PFTs, tests are completed the screening of respiratory infections and chest computed tomographic scan (CT-scan) is performed. A report from the National Institute of Health described the following criteria required for the diagnosis of BOS : FEV1/vital capacity < 0.7, FEV1 < 75% or a decline >/= 10% from baseline, residual volume > 120%, absence of documented infection, and the presence of CT-scan signs suggestive of BOS : air trapping by expiratory CT or small airway thickening or bronchiectasis.

BOS severity depends on the development of fibrotic and fixed damages, poorly responding to therapies. New tools are needed in order to favor early BOS diagnosis.

A recent study from our center showed that repeated CT-scans in stem cell transplant patients is associated with increased risk of neoplasia. In addition, recent studies from our center evaluated the use of pulmonary MRI providing good performance without X-ray exposure (Dournes G et al, Radiology 2015 et Dournes G et al, Eur Radiol 2015).

More recently, Renne et al (Radiology 2015) studied the performance of pulmonary MRI coupled with oxygen transfer analysis for the diagnosis of chronic lung allograft dysfunction. This study showed altered imaging parameters in patients developing BOS, including patients with early BOS stage (0p stage).

As pathogenic mechanisms seem to be shared between post-stem cell transplant and post-lung transplant BOS, we hypothesize that pulmonary MRI with oxygen transfer analysis and ultra short echo time may represent a non-invasive, non-irradiating and sensitive research tool for the detection and quantification of pulmonary lesions in patients screened for post-stem cell transplant BOS.

Thus, 20 patients who underwent allogeneic stem cell transplantation and show abnormal respiratory function over a 2 year period study are expected. They will be included according to the following criteria : age > 18 yo, > 3 months post-transplant, absence of documented pulmonary infection, or with a minimum of 6 weeks after a documented pulmonary infection, and the following BOS criteria : abnormal PFTs (FEV1/VC < 0.7, FEV1 < 0.75, residual volume < 120% of expected value) and/or chest CT-scan showing air trapping or small airway thickening. Similarly to lung transplant criteria, stage 0p BOS defined according to FEF25-75 values (Estenne et al, JHLT 2002), for which pulmonary MRI with oxygen transfer may guide to early BOS diagnosis, will be added.

Patients who give their consent will perform a pulmonary MRI, in the absence of contraindication, using different sequences to evaluate morphologic and functional performances of pulmonary MRI. We will compare CT-scan and MRI performances using blinded analysis from two radiologists.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 yo ;
* Patient who underwent an allogeneic stem cell transplantation (SCT)
* > 3 months post-SCT
* With evidence of

  * respiratory symptoms, and/or
  * Pathological PFTs defined by : obstructive syndrome (FEV1 :vital capacity/CVF < 0.7), FEV1 < 0.75 of pre-SCT values, residual volume > 120%, and/or ;
  * Altered PFTs consistent with 0p stage described in lung transplantation BOS: FEV1 decline ≥ 10 % and/or FEF25-75 decline ≥ 25% compared to pre-SCT PFTs, and/or ;
  * Abnormal chest CT-scan with findings consistent with BOS: evidence of air trapping on expiratory CT-scan, bronchiectasis, and/or airway thickening.

Exclusion Criteria:

* Contraindication for MRI ;
* Contraindication of oxygen administration ;
* Decompensation of altered respiratory function ;
* Acute respiratory infection (bacterial, fungal or viral) documented in the last 6 weeks ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
lung MRI concordance as compared to chest CT-scan | Baseline
  lung MRI concordance as compared to chest CT-scan for the description of morphological abnormalities necessary for the diagnosis of BOS after HSCT. It will be evaluated using lung MRI performed after inclusion (Baseline) using a standardized procedure. The agreement between MRI and chest CT-scan for the presence or absence of the following features, will be measured at the segmental level: airway thickening, bronchiectasis, air trapping.

SECONDARY OUTCOMES:
Bhalla Score precision in morphological MRI | Baseline
  Measure of Bhalla Score precision in morphological MRI for the diagnosis of post-transplant BOS
Bhalla Score in CT scan | Baseline
  Bhalla Score in CT scan
oxygen transfer capacity | Baseline
  Measure of oxygen transfer capacity (percentage of intra-pulmonary signal variation before and after inhalation of oxygen);
Force Expiratory Volume | Baseline
  Force Expiratory Volume (FEV, l)
FEV1/VC | Baseline
  FEV1/VC (Tiffeneau),
Residual volume | Baseline
  Residual volume (l)
total lung capacity | Baseline
  Total lung capacity (l)
BOS stages | Baseline
  BOS stages (0 : FEV1 > 90%, and FEF25-75 > 75% from baseline; 0p : 10-19% decrease in FEV1, and/or by a >/= 25% decrease in FEF 25-75 from baseline; 1: FEV1 60-79% ; 2: FEV1 40-59% ; 3: FEV1</= 39)
intra-observer repeatability of the Bhalla score in CT scan | Baseline
  Intraclass coefficient and Bland-Altman's test
intra-observer repeatability of the Bhalla score in MRI | Baseline
  Intraclass coefficient and Bland-Altman's test
intra-observer repeatability of the measure of oxygen transfer capacity | Baseline
  Intraclass coefficient and Bland-Altman's test
inter-observer reproducibility of the Bhalla score in CT scan | Baseline
  Intraclass coefficient and Bland-Altman's test
inter-observer reproducibility of the Bhalla score in MRI | Baseline
  Intraclass coefficient and Bland-Altman's test
inter-observer reproducibility of the measure of oxygen transfer capacity | Baseline
  Intraclass coefficient and Bland-Altman's test

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No